CLINICAL TRIAL: NCT01693237
Title: Feedback Versus no Feedback to Improve Patient Outcome in Group Psychotherapy for Eating Disorders: A Randomised Clinical Trial
Brief Title: Improving Patient Outcome in Group Therapy for Eating Disorders
Acronym: F-EAT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marianne Lau, MD, DSci. (Other Government)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Sponsor-Investigator, Marianne Lau, MD, DSci., Research Manager, Psychotherapeutic Center Stolpegard
Organization: Psychotherapeutic Center Stolpegard (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-084080
Record Dates: First submitted 2012-08-28; First posted 2012-09-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Bulimia Nervosa (BN); Binge Eating Disorder (BED); Eating Disorder Not Otherwise Specified (EDNOS)
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group psychotherapy (Active Comparator): 20 sessions of systemic and narrative group psychotherapy
  Interventions: Other: Group psychotherapy
- Group psychotherapy with feedback (Experimental): 20 sessions of systemic and narrative group psychotherapy with session-to-session feedback to patient and therapist.
  Interventions: Other: Group psychotherapy with feedback

INTERVENTIONS:
Other: Group psychotherapy — 20 sessions of systemic and narrative group therapy
  Arms: Group psychotherapy
Other: Group psychotherapy with feedback — 20 sessions of systemic and narrative group therapy
  Arms: Group psychotherapy with feedback

SUMMARY:
The current trial aims to investigate the impact of continuous feedback on dropout and outcome in group therapy. The hypothesis is that continuous feedback to patient and therapist on treatment progress and alliance will 1) increase adherence and 2) increase treatment outcome.

DETAILED DESCRIPTION:
Background: In the psychotherapy of eating disorders, a dropout rate between 30% and 50% is reported internationally. The fact that up to half of the patients drop out of treatment calls for ways to improve it. Research shows that feedback to patient and therapist increases outcome and reduces the number of dropouts; however there is only three published works on the effect of feedback in eating disorders treatment. Therefore, the present trial, at the eating disorders unit at Stolpegaard Psychotherapy Centre, Gentofte, Denmark, may contribute to necessary improvements in the field.

Objective: The current trial, which will be conducted from August 2012 to August 2014, aims to investigate the impact of continuous feedback on adherence and outcome in group psychotherapy. The hypothesis is that continuous feedback to patient and therapist on treatment progress and alliance will 1)increase adherence 2) increase treatment outcome.

Method: The trial is set up in a randomized design with 159 patients allocated to a) treatment with feedback intervention or b) treatment as usual.

Participants: The participants are diagnosed with Bulimia Nervosa, Binge Eating Disorder or Eating Disorder Not Otherwise Specified.

Interventions: In the experimental group, two sets of feedback measures are added to the standard treatment: Outcome Rating Scale (ORS) and Group Session Rating Scale (GSRS). The ORS assesses areas of life functioning known to change as a result of therapeutic intervention. The GSRS assesses key dimensions of effective therapeutic relationships.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older.
* BMI of minimum 20.
* Meet the diagnostic criteria for Bulimia Nervosa, Binge Eating Disorder or EDNOS according to DSM- IV.

Exclusion Criteria:

* Acute suicidal risk.
* Psychosis.
* Severe depression.
* Abuse of alcohol, medicine and/or narcotics up to 3 months before referral.
* Use of cannabis once a month is accepted at intake but must stop during treatment.
* Concomitant psychotherapeutic/ psychiatric treatment outside Stolpegaard Psychotherapy Centre.
* Severe or non-regulated physical co-morbidity.
* Pregnancy.
* Unable to understand Danish.
* Previous participation in the current trial.
* Considered unable to attend treatment sessions as planned.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Adherence | At end of treatment. Participants will be followed for the duration of treatment, an expected average of 20 weeks.
  Treatment adherence in the intervention period defined as a rate, i.e., number of attended therapy sessions divided by the number of planned therapy sessions. If a patient ends therapy prematurely, and this is in accordance with the therapists, the number of attended sessions will be set equal to the planned number of sessions.

SECONDARY OUTCOMES:
Eating Disorders Examination Interview | At intake, end of treatment and follow-up. Participants will be followed for the duration of treatment and follow-up, an expected average of 3 years.

OTHER OUTCOMES:
Self-Harm Inventory | At end of treatment? Participants will be followed for the duration of treatment, an expected average of 20 weeks.
Outcome Rating Scale | At start of treatment and during treatment. Participants will be followed for the duration of treatment, an expected average of 20 weeks.
Symptom Check List-90R | At start of treatment and during treatment. Participants will be followed for the duration of treatment, an expected average of three years.
Sheehan Disability Scale | At start of treatment and during treatment. Participants will be followed for the duration of treatment, an expected average of three years.
WHO-Five Well-being Index | At start of treatment and during treatment. Participants will be followed for the duration of treatment, an expected average of three years.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne E. Lau, D.Sci., Principal Investigator — Stolpegaard Psychotherapy Centre
Locations (1):
- Stolpegaard Psychotherapy Centre, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Davidsen AH, Poulsen S, Lindschou J, Winkel P, Trondarson MF, Waaddegaard M, Lau M. Feedback in group psychotherapy for eating disorders: A randomized clinical trial. J Consult Clin Psychol. 2017 May;85(5):484-494. doi: 10.1037/ccp0000173. Epub 2017 Mar 23. PMID 28333513
- [Derived] Davidsen AH, Poulsen S, Waaddegaard M, Lindschou J, Lau M. Feedback versus no feedback in improving patient outcome in group psychotherapy for eating disorders (F-EAT): protocol for a randomized clinical trial. Trials. 2014 Apr 23;15:138. doi: 10.1186/1745-6215-15-138. PMID 24754974
- See also: Stolpegaard Psychotherapy Centre — http://www.psykiatri-regionh.dk/menu/Centre/Psykiatriske+centre/Psykoterapeutisk+Center+Stolpegard/Forskning/F-EAT/Abstract/